CLINICAL TRIAL: NCT06149117
Title: A Single-center, Open-label, Randomized, Single-dose, Crossover Study to Compare the Equivalence of the Fasting Oral Test Formulation Azithromycin Capsule to Reference Formulation Sumamed *in Healthy Adult Chinese Subjects
Brief Title: Bioequivalence Study of Azithromycin Capsule and Reference Formulation Sumamed * in Healthy Adult Subjects in China
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Yi Fang, Professor of Pharmacy, Peking University People's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: I-2022-03
Record Dates: First submitted 2023-09-04; First posted 2023-11-28 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Upper Respiratory Tract Infection; Lower Respiratory Infection; Skin Infection; Subcutaneous Tissues Infection; Genital Infection
MeSH Terms: conditions — Respiratory Tract Infections; Cellulitis | interventions — Azithromycin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- test product (T) azithromycin capsule and reference product (R) azithromycin capsule "Sumamed®" (Experimental): TR
  Interventions: Drug: test product (T) azithromycin capsule and reference product (R) azithromycin capsule "Sumamed®"
- reference product (R) azithromycin capsule "Sumamed®"and test product (T) azithromycin capsule (Experimental): RT
  Interventions: Drug: test product (T) azithromycin capsule and reference product (R) azithromycin capsule "Sumamed®"

INTERVENTIONS:
Drug: test product (T) azithromycin capsule and reference product (R) azithromycin capsule "Sumamed®" — Take one capsule orally every cycle(T or R)

SUMMARY:
Main research purpose

To investigate the pharmacokinetics of the test preparation azithromycin capsule and the reference preparation azithromycin capsule (Sumamed®) in Chinese healthy adult subjects by single oral administration in fasting state, and to evaluate the bioequivalence of the two preparations by oral administration in fasting state.

Secondary research purpose

To investigate the safety of the test preparation azithromycin capsule and the reference preparation "Sumamed®" in healthy subjects.

DETAILED DESCRIPTION:
The fasting trial was designed with single-center, open, randomized, single-dose, two-cycle, two-sequence and cross-dosing trials.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet all of the following inclusion criteria to be enrolled in the study:

  1. Before the test, voluntarily sign informed consent, fully understand the test content, process and possible adverse reactions, and be able to complete the study in accordance with the requirements of the test plan;
  2. Chinese male and female subjects aged 18-45 years old (including 18 and 45 years old);
  3. The weight of male subjects is not less than 50.0kg, the weight of female subjects is not less than 45.0kg, the body mass index (BMI = weight/height 2 (kg/m2)), the body mass index is in the range of 19.0~26.0 kg/m2 (including the cut-off value).

Exclusion Criteria:

* One of the following conditions will be excluded:

  1. (Consultation, systematic inquiry) The study physician considers it inappropriate for participants to have past or present chronic or serious diseases of cardiovascular, liver, kidney, respiratory, blood and lymphatic, endocrine, immune, psychiatric, nervous, gastrointestinal, metabolic and skeletal systems;
  2. Clinically significant abnormalities judged by clinicians during the screening period, including physical examination, vital signs examination, electrocardiogram or clinical laboratory examination;
  3. (Check) male QTc interval greater than 450ms, female QTc interval greater than 470ms;
  4. (consultation) past or current epilepsy or a history of seizures;
  5. Patients with a history of cholestatic jaundice/hepatic insufficiency after previous use of azithromycin;
  6. (consultation) people who have a history of specific allergies (asthma, etc.) or are currently suffering from allergic diseases (urticaria, eczema, etc.), or are allergic to two or more drugs, foods such as milk or pollen, or are known to be allergic to components or analogizes of this drug (such as azithromycin, erythromycin, other macrolides or ketonolactones);
  7. (consultation) have dysphagia or any history of gastrointestinal diseases that affect drug absorption (such as stomach or small intestine resection, atrophic gastritis, gastrointestinal bleeding, obstruction, etc.);
  8. (consultation) patients with any disease that increases the risk of gastrointestinal bleeding (such as acute gastritis or gastric and duodenal ulcers);
  9. (consultation) Patients with venous blood collection difficulties and a history of fainting needles and fainting blood;
  10. (consultation, examination) female subjects who are in pregnancy, breastfeeding or pregnancy test results are positive;
  11. (Consultation) Subjects (including male subjects) who have not taken effective contraception within 14 days before the first dose, or who have a pregnancy, sperm donation or egg donation plan within 6 months after the last dose, see Appendix 2 for specific contraceptive methods;
  12. (examination) Human immunodeficiency virus antibody (screening), hepatitis B virus surface antigen test, hepatitis C virus antibody test, treponema pallidum antibody any test result is positive;
  13. (consultation, examination) have a history of drug abuse within five years, or have used drugs within 3 months before screening, or urine drug screening positive;
  14. (consultation, examination) those who consumed an average of more than 14 units of alcohol per week (1 unit =360 mL beer or 45 mL liquor with 40% alcohol or 150 mL wine) in the three months prior to screening, or those who could not stop alcohol intake from 24 hours before medication to the completion of the blood sample collection for that cycle, or those who tested positive for alcohol breath;
  15. (Consultation) Those who smoked more than 5 cigarettes per day on average in the 3 months before screening or used e-cigarette products or refused to stop smoking (including e-cigarettes) during check-in;
  16. (Consultation) patients with surgery or severe trauma that the investigator determined would affect drug absorption, distribution, metabolism, or excretion, or who are scheduled to be hospitalized for surgery, dental surgery, or hospitalization during the study period;
  17. Blood donation and/or component blood within 3 months before screening or planned blood donation and/or component blood during the test period, or large blood loss (>400mL, except for female physiological blood loss), or blood transfusion or use of blood products;
  18. Patients who have participated in any drug clinical trials and used drugs within 3 months before screening (consultation);
  19. (Consultation) Those who have taken any drug that alters liver enzyme activity or interacts with azithromycin (such as antacids, ergotamine or dihydroergotamine, fluconazole, efavirenz, nefinavir, etc.) within 28 days before the first dose;
  20. (Consultation) Those who have taken any prescription drugs (including vaccines) within 14 days before the first dose;
  21. (Consultation) Those who have taken any non-prescription drugs, Chinese herbs or health products for the prevention and/or treatment of their own diseases within 14 days prior to the first medication;
  22. (Consultation) 48 hours before the first dose until the end of the study, those who cannot avoid eating a special diet (such as grapefruit and products containing grapefruit components) or have vigorous exercise, or have other factors affecting drug absorption, distribution, metabolism, excretion, etc.;
  23. (Consultation) patients who cannot avoid consuming any food or drink rich in caffeine or xanthines (such as coffee, tea, chocolate, cocoa, milk tea, etc.) 48 hours before taking the drug until the end of the study;
  24. Subjects deemed unsuitable by other investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-11-16 (Actual); Primary Completion 2023-04-03 (Actual); Study Completion 2023-04-03 (Actual)

PRIMARY OUTCOMES:
Cmax | Pre-dose and after dose 7 days
  PK parameters comparison between test product azithromycin capsuleand Sumamed®: Cmax
AUC0-t | Pre-dose and after dose 7 days
  PK parameters comparison between test product azithromycin capsuleand Sumamed®:AUC0-t
AUC0-∞ | Pre-dose and after dose 7 days
  PK parameters comparison between test product azithromycin capsuleand Sumamed®:AUC0-∞

SECONDARY OUTCOMES:
Tmax | Pre-dose and after dose 7 days
  PK parameters comparison between test product azithromycin capsuleand Sumamed®:Tmax
t1/2 | Pre-dose and after dose 7 days
  PK parameters comparison between test product azithromycin capsuleand Sumamed®:t1/2
λz | Pre-dose and after dose 7 days
  PK parameters comparison between test product azithromycin capsuleand Sumamed®:λz
AUC_%Extrap | Pre-dose and after dose 7 days
  PK parameters comparison between test product azithromycin capsuleand Sumamed®:AUC_%Extrap

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China